CLINICAL TRIAL: NCT04647305
Title: Effectiveness and Adherence to Closed Face Shields to Prevent COVID-19 Transmission: A Randomized Controlled Trial
Brief Title: Effectiveness and Adherence to Closed Face Shields to Prevent COVID-19 Transmission
Acronym: COVPROSHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: United Nations (Other)
Responsible Party: Principal Investigator, Andrea Ramirez Varela, Assistant Professor of Epidemiology, University of Los Andes, Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1010166518
Record Dates: First submitted 2020-11-24; First posted 2020-11-30 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV-2 Infection
Keywords: Face shield; Visor; Adherence; Prevention; COVID-19; SARS-CoV-2 infection; Controlled Clinical Trial; Seroprevalence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed face shield + Surgical face mask (Experimental): Each participant will wear 21 surgical face masks corresponding to the follow-up days in the randomized clinical trial, as well as one closed face shield. Additionally, each participant will receive an educational intervention (video).
  Interventions: Other: Closed face shield with Surgical face mask use
- Surgical face mask (Active Comparator): Each participant will wear 21 surgical face masks corresponding to the follow-up days in the randomized clinical trial. Additionally, each participant will receive an educational intervention (video).
  Interventions: Other: Surgical face mask use only

INTERVENTIONS:
Other: Closed face shield with Surgical face mask use — Use of a closed face shield with a surgical face mask during daily activities. The educational intervention will provide recommendations on COVID-19 prevention and proper use of the closed face shield and the surgical face masks.
  Arms: Closed face shield + Surgical face mask
Other: Surgical face mask use only — Use of a surgical face mask during daily activities. The educational intervention will provide recommendations on COVID-19 prevention and the proper use of surgical face masks.
  Arms: Surgical face mask

SUMMARY:
A non-inferiority randomized controlled trial that aims to determine the effectiveness and adherence of the use of closed-face shields and surgical face masks in comparison with the use of surgical face masks for the prevention of SARS-CoV-2 infection in working adults in the city of Bogota, Colombia.

DETAILED DESCRIPTION:
Introduction

According to the Johns Hopkins University coronavirus resource center, COVID-19 has caused more than 1,399,373 deaths globally (as of November 24, 2020), and more than 59 million cases have been reported worldwide. Governments have been forced to establish various preventive measures to control transmission in the communities. The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is transmitted among close contacts mainly via respiratory droplets generated when an infected person coughs or sneezes. Likewise, airborne transmission through fomites/aerosols have been described due to the persistence of SARS-CoV-2 on different surfaces and the environment. SARS-CoV-2 causes the coronavirus disease 2019 (COVID-19), the respiratory illness responsible for the ongoing COVID-19 pandemic.

Physical distancing, face mask use, and eye protection had affected stopping SARS-CoV-2 transmission. While there is evidence of the use of face masks as a strategy to control respiratory infections and prevent the inhalation of large droplets and sprays, there is a need to determine the effectiveness of closed-face shields to prevent transmission in community settings. Despite the available reports, none of the randomized clinical trials have been conducted in the community setting. Although scarce, there is promising evidence showing that using face shields may bring an extra benefit in protecting airborne diseases, like COVID-19. Face shields have the benefits of preventing constant contact between face and hands, preventing airflow with possible infected particles from reaching the face, and protecting the eyes.

As of November 24, 2020, more than 1,254,979 cases have been reported in Colombia, and more than 35,479 deaths have occurred (a fatality rate of 2.83%). So far, no massive seroprevalence studies have been carried out in Colombia, that would determine the presence of Immunoglobulin G (IgG) and Immunoglobulin M (IgM) anti-SARS-CoV-2 antibodies, therefore, the level of immunity of the population and the likelihood of further waves of the disease. The first study to determine seroprevalence in Colombia found that, in a sample of 1368 people on the Caribbean coast of Colombia, 55.3% of the participants had anti-SARS-CoV-2 antibodies. The study of seroprevalence that is currently implemented by the Colombian National Institute of Health has not yet yielded results. Bogota, the country's capital district, has the highest number of confirmed cases compared to other departments and cities, but no studies have been conducted to determine what is level of immunity in the city´s population.

Therefore, epidemiological surveillance strategies are carried out to identify asymptomatic and symptomatic patients, trace contacts, and isolate cases to break transmission chains. As a result, an initiative called the CoVIDA project, which enrolls several institutions from academia to hospitals and the health authorities has emerged to support the epidemiological surveillance system of the city. This strategy is based on reverse transcription polymerase chain reaction (RT-PCR) testing for SARS-Cov-2 detection in populations that, because of their work and high mobility in public places, are at high risk of infection and spread of the virus and has contributed to inform the health authorities and help them in the effective decision-making for public policy management.

The CoVIDA project is a study that follows up participants for 21 days and has enrolled more than 33,667 participants since April 2020. The study has included participants whose occupations have high mobility in the community, such as police, military, firefighters, private and public service drivers, shopkeepers, domiciliary, and private security guards, among others. Participants are mostly between 30 and 39 years old, followed by 20 to 29 years old, and there is a lower proportion of the elder population. As of November 24, 2020, from the total of 33,667 participants included in this epidemiological surveillance, 4.35% presented a positive result for the SARS -CoV-2 RT-PCR test.

The present non-inferiority randomized controlled trial aims to determine the effectiveness and adherence of closed face shields plus face mask use compared to face mask use only to prevent SARS -CoV-2 transmission in working adults of Bogota, Colombia.

Methods

Non-inferiority randomized controlled trial nested within a cohort, with a parallel design of 1:1 allocation ratio. Study participants will be recruited through the CoVIDA project that enrolls working adults in Bogota as part of the COVID-19 epidemiologic surveillance. Those who consent to participate in the trial will be randomized for a group wearing closed face shield plus face masks or a group wearing face masks only. Participants will also receive an educational intervention about COVID-19 prevention and the proper use of face shields and face masks. The intervention will last 21 days and includes a COVID-19 symptoms report and verification of protective elements use (adherence). The RT-PCR test and antibody test will be repeated on day 21. A total sample size of 194 participants, 97 per arm, is required to be 80% sure that the upper limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will exclude a difference in favor of the standard group of more than 5%. If 20% of rejects or losses to follow-up are considered, 233 will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Negative RT-PCR test at the beginning of the study.
* Negative SARS-CoV-2 serological Elecsys Anti-Sars-CoV-2 test at the beginning of the study.
* Living in a geographic area with active COVID-19 transmission (number of
* cases reported locally).
* Living in a geographic area that has been determined by the Colombian National Statistics Department (DANE) to have a medium, medium-high, and high vulnerability index (higher prevalence of comorbidities and social and economic vulnerabilities.
* Working outside the home for at least two days a week, during the last week.
* Acceptance to participate in the study regardless of the trial arm assignment through verbal informed consent.

Exclusion Criteria:

* Retired adults or unemployed
* Adults referring previous diagnosis of COVID-19 confirmed by RT-PCR tests or serological antibody tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
COVID-19 incidence | 21 days of follow-up, RT-PCR test at day 21
  The numerator will be the number of cases or the number of persons with laboratory evidence of present infection. In this case, a person with a positive result of a RT-PCR test for SARS-CoV-2 detection. The denominator will be the number of persons allocated in the determined group. Incidence of SARS-CoV-2 infection has been used as a risk measure in several studies, in which comparison groups are made. This risk measure will also allow the calculation of association measures such as RR (relative risk) in both intervention groups.

SECONDARY OUTCOMES:
Adherence to closed face shields use | 21 days of follow-up
  Adherence to closed face shields is defined as proper daily use of this protective element, which must be worn daily outside the home, and never touch the facial area of the protector. Face shields must be washed daily. Additionally, adherence to face masks is defined as a proper daily use which consists of wearing it covering the nose and mouth, as well as throwing it away daily. A questionnaire intended to evaluate the frequency of use and perception about the advantages of closed face shields and face mask use, as well as the barriers of their use, will be implemented in the participants at the end of the follow-up period.
Percentage of participants with a positive serological test at baseline | Serological test at day 1
  It will be calculated as the number of participants with a positive serological test over the total of people eligible for the clinical trial at baseline.
Percentage of seroconversion in the experimental group and active control group | Serological test at day 21.
  The numerator will be the number of individuals in each group with a positive serological test at end of the study, and the denominator will be the total number of participants assigned to each group.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Pacheco Gurruchaga, MSc, Principal Investigator — United Nations; Juan D. Martin, MSc, Principal Investigator — United Nations; Luis J. Hernandez Florez, PhD, Study Chair — University of Los Andes, School of Medicine; Juan J. Yepes Nuñez, PhD, Study Chair — University of Los Andes, School of Medicine; Giancarlo Buitrago Gutierrez, PhD, Principal Investigator — University of Los Andes; Rachid Laajaj, PhD, Principal Investigator — University of Los Andes; Eduardo Behrentz, PhD, Study Director — University of Los Andes; José D. Pinzón, MSc, Principal Investigator — Pontificia Universidad Javeriana; Jhon M. Gonzalez, PhD, Principal Investigator — University of Los Andes, School of Medicine; Silvia Restrepo Restrepo, PhD, Principal Investigator — University of Los Andes
Locations (1):
- Universidad de los Andes, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
After publication of main results, data will be available for other researchers such as: Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: A formal request sent to the principal investigator.

REFERENCES:
- [Derived] Varela AR, Gurruchaga AP, Restrepo SR, Martin JD, Landazabal YDC, Tamayo-Cabeza G, Contreras-Arrieta S, Caballero-Diaz Y, Florez LJH, Gonzalez JM, Santos-Barbosa JC, Pinzon JD, Yepes-Nunez JJ, Laajaj R, Buitrago Gutierrez G, Florez MV, Fuentes Castillo J, Quinche Vargas G, Casas A, Medina A, Behrentz E; CoVIDA Working Group. Effectiveness and adherence to closed face shields in the prevention of COVID-19 transmission: a non-inferiority randomized controlled trial in a middle-income setting (COVPROSHIELD). Trials. 2022 Aug 20;23(1):698. doi: 10.1186/s13063-022-06606-0. PMID 35987694
- [Derived] Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, Engela-Volker JS, McElvenny D, Rhodes S, Stocking K, Fletcher T, Martin C, Noertjojo K, Sampson O, Verbeek JH, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2022 May 6;5(5):CD015112. doi: 10.1002/14651858.CD015112.pub2. PMID 35514111